CLINICAL TRIAL: NCT04529655
Title: Digital Capillary Refill for Monitoring of Sepsis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dr. David Sheridan, Assistant Professor of Emergency Medicine, Oregon Health and Science University
Other Study IDs: STUDY00021286
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sepsis: Patients admitted to the ICU with sepsis will be enrolled and monitored at time sequential time points during their treatment
  Interventions: Device: Capillary Refill Assessment

INTERVENTIONS:
Device: Capillary Refill Assessment — Device to quantify capillary refill time

SUMMARY:
Observational study for monitoring of capillary refill time in sepsis

DETAILED DESCRIPTION:
This is an observational studying assessing changes in capillary refill time over the course of sepsis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical evidence of a known or suspected infection and orders written for administration of IV antibiotics
2. Hypotension as defined by the need for any vasopressor (and 1 liter of fluid already administered) OR respiratory failure defined by assisted ventilation (includes mechanical ventilation and BIPAP), CPAP, or greater than or equal to 6 liters/minute of supplemental oxygen

Exclusion Criteria:

1. No consent/inability to obtain consent from the participant or a legally authorized representative
2. Diagnosis of cirrhosis by medical chart review
3. Liver transplant recipient
4. AST or ALT greater than five times upper limit of normal
5. Diagnosis of ongoing chronic alcohol use disorder/abuse by chart review; if medical record unclear, use Appendix F
6. Clinical diagnosis of diabetic ketoacidosis or other condition such as profound hypoglycemia that requires hourly blood glucose monitoring
7. Hypersensitivity to Acetaminophen or Vitamin C
8. Patient, surrogate or physician not committed to full support (Exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
9. Home assisted ventilation (via tracheotomy or noninvasive) except for CPAP/BIPAP used only for sleep-disordered breathing
10. Current active kidney stone
11. Known history of oxalate kidney stones or history of oxalate nephropathy
12. Kidney transplant recipient
13. Use of home oxygen for chronic cardiopulmonary disease
14. Moribund patient not expected to survive 24 hours
15. Underlying malignancy or other condition with estimated life expectancy of less than 1 month
16. Pregnant woman, woman of childbearing potential without a documented negative urine or serum pregnancy test during the current hospitalization, or woman who is breast feeding
17. Prisoner
18. Enrollment in another critical care based pharmacologic interventional trial
19. Treating team unwilling to enroll because of intended use of Acetaminophen or Vitamin C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the ICU, ED or inpatient floor with sepsis defined as a concern for an infection with either hemodynamic or respiratory organ failure on intravenous antibiotics will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Blood lactate Level | during procedure
  Correlation of Capillary refill to blood lactate

SECONDARY OUTCOMES:
Vasoactive | 24 hours
  Correlation of capillary refill to need for vasoactive medications
28 day hospital mortality | 28 days
  Correlation of initial capillary refill time to 28 day hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: David Sheridan, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No